CLINICAL TRIAL: NCT03681808
Title: A Study to Evaluate the Safety and Effectiveness of the Biotrue ONEday for Astigmatism Soft Contact Lens When Worn on a Daily Basis
Brief Title: Evaluate the Safety and Effectiveness of the Biotrue ONEday for Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 885
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: Investigator/Sponsor masked, randomized, open-label, parallel-group, multicenter study
Who Masked: Investigator
Masking Description: Subjects will be dispensed product according to the treatment arm corresponding to their randomization and will be unmasked. The Investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test (Experimental): Soft Contact Lens
  Interventions: Device: Test
- Control (Active Comparator): Contact lens
  Interventions: Device: Control

INTERVENTIONS:
Device: Control — Contact Lens
  Arms: Control
Device: Test — Soft Contact Lens
  Arms: Test

SUMMARY:
Comparing Test Lens for Astigmatism Soft Contact Lens (Test) to 1-Day Control for Astigmatism contact lenses (Control).

DETAILED DESCRIPTION:
This is a multicenter, randomized 1:1, parallel-group, bilateral, Investigator-masked study at 13 investigative sites in the United States (US) in a population including Chinese subjects (maternal and paternal grandparents born in China)

ELIGIBILITY:
Inclusion Criteria:

* Subject must be of legal age (at least 18 or as defined by state law) on the date the ICF is signed and have the capacity to provide voluntary informed consent.
* Subject must be able to read, understand and provide written informed consent on the IRB approved ICF and provide authorization as appropriate for local privacy regulations.
* Subject must have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings (greater than Grade 1 and/or presence of infiltrates) and have clear central 6 mm corneas.
* Subject must be an adapted wearer of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.

Exclusion Criteria:

* Subject has worn gas permeable (GP) contact lenses within last 30 days or polymethylmethacrylate (PMMA) lenses within last 3 months.
* Subject has systemic disease affecting ocular health.
* Subject is using any systemic or topical medications that will affect ocular physiology or lens performance.
* Subject has an active ocular disease (for example but not limited to papillary conjunctivitis, any conjunctivitis: viral, bacterial, allergic), any corneal infiltrative response or are using any ocular medications.
* Subject has any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Companies
Locations (13):
- United States (13):
  - Bausch Site 117, Irvine, California
  - Bausch Site 107, San Diego, California
  - Bausch Site 101, San Francisco, California
  - Bausch Site 108, San Jose, California
  - Bausch Site 104, Sunnyvale, California
  - Bausch Site 102, Jacksonville, Florida
  - Bausch Site 116, Bloomington, Illinois
  - Bausch Site 110, Brighton, New York
  - Bausch Site 118, New York, New York
  - Bausch Site 111, New York, New York
  - Bausch Site 114, Raleigh, North Carolina
  - Bausch Site 105, Houston, Texas
  - Bausch Site 115, Issaquah, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Biotrue: Biotrue ONEday for Astigmatism Soft Contact Lens®
- Acuvue: 1-Day Acuvue Moist for Astigmatism Contact Lens
Period: Overall Study
Arm/Group | Biotrue | Acuvue
Started | 123 | 119
Completed | 109 | 102
Not Completed | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biotrue | Acuvue | Total
Number analyzed (Participants) | 123 | 119 | 242
Age, Continuous [Mean (Full Range); unit: years] | 33.7 [19 to 59] | 32.9 [18 to 71] | 33.3 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 72 | 150
  Male | 45 | 47 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 60 | 59 | 119
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 16 | 8 | 24
  White | 42 | 49 | 91
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 1
Ancestry [Count of Participants; unit: Participants]
  Chinese | 45 | 41 | 86
  Non-Chinese | 78 | 78 | 156

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving a Contact Lens Corrected Distance logMAR VA of 0.04 or Better
Description: The proportion of participants achieving a contact lens corrected distance logMAR VA of 0.04 or better in both eyes
Time Frame: Evaluated at the 1 week follow up visit
Population: The Per Protocol (PP) Population included all randomized participants without major protocol deviations who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Biotrue | Acuvue
Number analyzed (Participants) | 106 | 98
Participants | 105 | 92

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Biotrue | Acuvue
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/119
Other Adverse Events (participants affected / at risk) | 0/123 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT03681808/Prot_SAP_000.pdf